CLINICAL TRIAL: NCT05024175
Title: Long-term Follow-up of Subjects Treated With CAR T Cells
Status: Recruiting | Type: Observational
Sponsor: Marcela V. Maus, M.D.,Ph.D. (Other)
Responsible Party: Sponsor-Investigator, Marcela V. Maus, M.D.,Ph.D., Sponsor Investigator, Massachusetts General Hospital
Organization: Massachusetts General Hospital (Other)
Other Study IDs: 20-721
Record Dates: First submitted 2021-08-23; First posted 2021-08-27 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-09

CONDITIONS: Long Term Adverse Effects; CAR-T; Duty to Follow Up; Adult; Progression-Free Survival; Disease-Free Survival; Overall Survival
Keywords: Long-Term Follow-up to CAR-T Cells; Follow-up Studies
MeSH Terms: conditions — Long Term Adverse Effects | interventions — Hematologic Tests

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- CAR T cells: * Eligibility to participate on this study if enrolled on a DF/HCC IRB corresponding main study and received infusion of CAR T cells
  * The research study procedures include evaluations and follow up visits: Timepoints of each evaluation and follow up visit- per protocol
  * Medical History/Physical Exam
  * Blood Test
  * Assessment of Disease: CT (Computerized Tomography) scan or PET-CT (Positron Emission Tomography-Computerized Tomography) scans.
  * Tumor biopsy.
  * Data Collection
  * Biobanking
  Interventions: Diagnostic Test: Disease assessments; Procedure: Tumor Biopsy; Diagnostic Test: Blood test

INTERVENTIONS:
Diagnostic Test: Disease assessments — CT (Computerized Tomography) scan or PET-CT (Positron Emission Tomography-Computerized Tomography) scans as per protocol
Procedure: Tumor Biopsy — Tumor Biopsy per protocol
Diagnostic Test: Blood test — Blood Test per protocol

SUMMARY:
This is a single site, non-randomized, open-label, long-term safety and efficacy follow-up study for Phase 1 studies that evaluate the safety and efficacy of CAR T cells: NCT05660369 (DF/HCC# 22-175) and NCT06026319 (DF/HCC# 23-474).

DETAILED DESCRIPTION:
This is a long-term safety and efficacy follow-up study for subjects who have been treated with CAR T cells in corresponding Phase I main studies that evaluated the safety and efficacy of CAR T cells in subjects.

No investigational treatment will be administered in this study.

The FDA (2020) recommends long-term follow up for subjects treated with gene therapy drug products to monitor for delayed adverse events (AEs), as well as durability of clinical response.

Therefore, after monitoring of subjects in the main studies has been completed (24 months after CAR T cells infusion, or <24 months after CAR T cells infusion if subject terminated early due to disease progression or due to discontinuing corresponding main study for any reason), subjects will be asked to participate in a long-term follow-up study (LTFU).

Subjects will be followed for up to 15 years following their last CAR T cells infusion in the corresponding main study.

ELIGIBILITY:
Inclusion Criteria:

Subjects will be asked to participate leading up to the last DF/HCC corresponding main study visit.

Subjects meeting the following criteria are eligible for study participation:

* Provision of voluntary written informed consent by subject
* CAR T cells were administered in DF/HCC IRB corresponding main study

Exclusion Criteria:

Subjects meeting the following criterion are to be excluded from study participation:

- Subject unable to comply with study requirements

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects will be asked to participate leading up to the last DF/HCC corresponding main study visit
Sampling Method: Non-Probability Sample
Enrollment: 45 (Estimated)
Dates: Start 2023-08-07 (Actual); Primary Completion 2038-08-01 (Estimated); Study Completion 2039-08-01 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | 1 month
  defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive
Overall Survival | 6 months
  defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive
Overall Survival | 12 months
  defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive
Overall Survival | 24 months
  defined as the time from randomization (or registration) to death due to any cause, or censored at date last known alive
Progresison Free Survival | 1 month
  PFS is defined as the number of days from the day of CAR T cells treatment to the first documented disease progression or date of death, whichever occurs first. Patients who are lost to follow up without a known date of progression or death due to any cause will be censored in the analysis at the date of their last available tumor assessment.
Progresison Free Survival | 6 months
  PFS is defined as the number of days from the day of CAR T cells treatment to the first documented disease progression or date of death, whichever occurs first. Patients who are lost to follow up without a known date of progression or death due to any cause will be censored in the analysis at the date of their last available tumor assessment.
Progresison Free Survival | 12 months
  PFS is defined as the number of days from the day of CAR T cells treatment to the first documented disease progression or date of death, whichever occurs first. Patients who are lost to follow up without a known date of progression or death due to any cause will be censored in the analysis at the date of their last available tumor assessment.
Progresison Free Survival | 24 months
  PFS is defined as the number of days from the day of CAR T cells treatment to the first documented disease progression or date of death, whichever occurs first. Patients who are lost to follow up without a known date of progression or death due to any cause will be censored in the analysis at the date of their last available tumor assessment.
New incidence or exacerbation of a pre-existing neurologic disorder or prior rheumatologic or other autoimmune disorder | Up to 15 Years
  An annual physical exam will be conducted for surveillance of manifestations indicative of oncoretroviral diseases.
New incidence of a hematologic disorder | up to 15 years
  An annual physical exam will be conducted for surveillance of manifestations indicative of oncoretroviral diseases.
Number of Participants with Treatment-Related Adverse Events as Assessed by CTCAE v 5.0 | up to 15 years
  NCI Common Terminology Criteria for Adverse Events (CTCAE)
Vector-derived RCL | baseline and in 3 months, 6 months, and annually up to 15 years
  Archiving of samples for potential detection of vector-derived RCL. RCL testing will be monitored at the central RCL lab (Indiana University) by a suitable qPCR assay for detection of the lentiviral vector (VSV-g DNA).
Assessment of CAR T cells persistence by VCN in peripheral blood | baseline and in 3 months, 6 months, every 6 months up to 5 years, and annually up to 15 years
  VCN will be performed in DNA from whole blood to monitor for persistence of vector sequence
Progression-free Survival | From post-CAR T cells infusion date until date of first documented disease progression or date of death from any cause, assessed up to 15 years post treatment
  The number of days from the day of CAR T cells treatment to the first documented disease progression or date of death, whichever occurs first. Patients who are lost to follow up without a known date of progression or death due to any cause will be censored in the analysis at the date of their last available tumor assessment.
Overall Survival | From post-CAR T cells infusion date until documented date of death from any cause, assessed post treatment every 6 months through 5 years and then annually up to 15 years
  The time from post-CAR T cells infusion to the date of death.

CONTACTS AND LOCATIONS:
Overall Officials: Matthew J Frigault, MD, Principal Investigator — Massachusetts General Hospital
Locations (1):
- Massachusetts General Hospital, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: Yes
The Dana-Farber / Harvard Cancer Center encourages and supports the responsible and ethical sharing of data from clinical trials. De-identified participant data from the final research dataset used in the published manuscript may only be shared under the terms of a Data Use Agreement. Requests may be directed to Sponsor Investigator or designee. The protocol and statistical analysis plan will be made available on Clinicaltrials.gov only as required by federal regulation or as a condition of awards and agreements supporting the research.
Supporting Information: Study Protocol, SAP
Time Frame: Data can be shared no earlier than 1 year following the date of publication
Access Criteria: Contact the Partners Innovations team at http://www.partners.org/innovation